CLINICAL TRIAL: NCT07142252
Title: Rezpegaldesleukin (NKTR-358) in New Onset Type 1 Diabetes Mellitus
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TN36 Rezpeg in New Onset
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: TrialNet; T1D
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: This trial will enroll 66 participants who will be randomly assigned in a 2:1 allocation to the following treatment arms:
  * Approximately 44 participants will be randomized to rezpegaldesleukin
  * Approximately 22 participants will be randomized to placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The randomization method will be stratified by TrialNet study site. The participants will not be informed regarding the intervention assignment until the end of the study. The investigator and clinic personnel will also be masked as to study assignment. Laboratories performing assays for this protocol will be masked as to the identity of biological material to be studied.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- rezpegaldesleukin (Experimental): Rezpegaldesleukin will be dosed at 12 μg/kg for subcutaneous injection. Rezpegaldesleukin will be provided as a 1.5 mg/mL sterile solution in a vial for injection preparation.
  Interventions: Drug: Rezpegaldesleukin
- Placebo (Placebo Comparator): The placebo dosing solution will be sterile saline for injection. The placebo will be administered in the same volume as the active comparator to maintain treatment masking.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rezpegaldesleukin — Rezpegaldesleukin will be dosed at 12 μg/kg for subcutaneous injection. Rezpegaldesleukin will be provided as a 1.5 mg/mL sterile solution in a vial for injection preparation. Study agent injections will be administered in the abdomen, back of the upper arm or the upper thigh of the participant.
  Other Names: NKTR-358
  Arms: rezpegaldesleukin
Drug: Placebo — Sterile saline for injection. Placebo will be administered in the same volume and as the active comparator to maintain treatment masking.
  Arms: Placebo

SUMMARY:
This Phase 2 study is a 2-arm, multi-center, double-masked, placebo-controlled, 2:1 randomized sequential trial design in new onset T1D participants (within 100 days of diagnosis). Participants will be administered rezpegaldesleukin/placebo once every 14 days over 26 weeks with an additional 6-month follow-up period.

DETAILED DESCRIPTION:
This protocol will enroll 66 participants within 100 days of T1D diagnosis who will be treated with either rezpegaldesleukin or placebo with subcutaneous injections over 26 weeks, administered once every 14 days. The rezpegaldesleukin/placebo treatment will be administered at the study site. Mixed meal tolerance testing will be done at the screening, baseline visit (V0) and at 3, 6 and 12 months during the study. Once the 26-week treatment period has been completed, participants will continue follow-up visits until 12 months from the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent or assent as appropriate and if < 18 years of age have a parent or legal guardian provide informed consent.
* Age ≥ 8 and ≤ 45 years at the time of signing informed consent and (as applicable) assent A.
* Diagnosis of T1D within 100 days of randomization.
* Positive for at least one islet cell autoantibody; GAD65A, mIAA (if obtained within 10 days of the onset of insulin therapy), IA-2A, ICA, or ZnT8A.
* Stimulated C-peptide of ≥ 0.2 pmol/mL measured during MMTT conducted at least 21 days from diagnosis of diabetes.
* Participants ≥ 18 years old to have body weight ≥ 35 kg and ≤ 130kg.
* Participants < 18 years old to have body weight > 5th and <98th percentile for age and sex.
* Willing to comply with intensive diabetes management.
* All CMV and/or EBV seronegative participants must be CMV and EBV PCR negative within 30 days of randomization and may not have had signs or symptoms of a CMV or EBV-compatible illness lasting longer than 7 days within 30 days of randomization.
* All CMV seropositive participants must be CMV PCR negative and all EBV seropositive participants must have a EBV PCR viral load < 2,000 IU/mL within 30 days of randomization. All participants may not have had signs or symptoms of a CMV or EBV-compatible illness lasting longer than 7 days within 30 days of randomization.
* Must meet "TrialNet Eligibility Minimum Immunization Recommendations" found in Appendix A of the MOO B.
* Be at least 4 weeks from last live vaccination prior to randomization.
* Participants that are not already immunized against the current year's influenza are required to receive non-live influenza vaccination at least 2 weeks prior to randomization when vaccine for the current or upcoming flu season is available.
* Be willing to forgo vaccines (other than killed influenza and COVID-19) during the treatment phase and the 3 months after study drug treatment period.
* If a female participant with reproductive potential, must be willing to avoid pregnancy (abstinence or highly effective contraceptive method) through the completion of the study and undergo pregnancy testing prior to each study visit.
* Males of reproductive age must use an adequate contraceptive method during the treatment phase and for 3 months following the last dose of study drug.

A Only adult participants ≥ 18 years old are permitted to be included in the first 18 enrolled participants in this study. Participants ≥ 12 and < 18 years of age are only permitted to screen for this study if the safety review of the first 18 adult participants is assessed favorably by the TrialNet DSMB in consultation with Nektar Safety Group. Once an additional 17 participants ages 12 to 45, including at least 9 participants aged 12-17, enroll and complete through the 6-month visit and have the safety review assessed favorably by the TrialNet DSMB in consultation with Nektar Safety Group, then the trial is permitted to screen and enroll the remaining 31 enrollees ≥ 8 and ≤ 45 years old. If data at either juncture do not support expansion into the pediatric ages, the trial will enroll the remaining participants to reach the target sample size with the currently approved age thresholds. See protocol sections 2.5 and 3.5 for additional details.

B For COVID-19 vaccination and HPV vaccination, all participants will be strongly encouraged to be up to date with COVID-19 vaccine(s) as indicated by country-specific guidelines and HPV vaccine(s) at least 2 weeks prior to randomization.

Exclusion Criteria:

* One or more screening laboratory values as stated

  * Neutrophils < 1,500 /μL
  * Lymphocytes < 800 /μL
  * Platelets < 100,000 /μL
  * Hemoglobin < 6.2 mmol/L (10.0 g/dL)
  * Eosinophils > 1,000 /μL
  * Potassium > 5.5 mmol/L or < 3.0 mmol/L
  * Sodium > 150 mmol/L or < 130 mmol/L
  * Estimated Glomerular Filtration Rate (eGFR) < 60 mL/min/1.73m2
  * AST or ALT or ALP > 2 times the upper limit of normal based on lab reference range
  * Total Bilirubin ≥ 1.5 times upper limit of normal unless diagnosed with Gilbert's syndrome
  * Serum creatinine > 2 times the upper limit of normal
* Current or ongoing use of non-insulin pharmaceuticals that affect glycemia within 7 days of the screening visit or any prohibited concomitant medication as listed in section 3.7.
* Concurrent treatment with systemic immunosuppressive agents (including biologics or steroids) - intranasal and inhaled corticosteroids are permitted as well as eye and ear drops containing corticosteroids.
* Have active signs or symptoms of acute infection at the time of randomization.
* Active acute or chronic infection requiring medical treatment (antibiotics, antiviral, antifungal) within 4 weeks of baseline visit unless approved by the Infectious Disease Committee.
* Have evidence of prior or current tuberculosis infection as assessed by Purified Protein Derivative (PPD), interferon gamma release assay (IGRA) or by history.
* Any present malignancies or history of malignancy within the past 5 years, other than a successfully treated nonmelanoma skin cancer.
* Be currently pregnant or lactating or anticipate becoming pregnant during the study.
* History of severe cardiac disease (i.e. myocardial infarction, unstable ischemic heart disease, cerebrovascular accident, stroke, stage 3 or 4 heart failure).
* Have evidence of current or past HIV or Hepatitis B infection.
* Have evidence of active Hepatitis C infection.
* History of organ allograft.
* Hypersensitivity to IL-2, PEG, or any components of the active drug.
* Had major surgery within 12 weeks before the screening visit or anticipates requiring major surgery during the study.
* Has any autoimmune disease other than T1D, stable thyroid, stable asthma, inactive Graves' disease or celiac disease (e.g., rheumatoid arthritis, polyarticular juvenile idiopathic arthritis, psoriatic arthritis, ankylosing spondylitis, multiple sclerosis, systemic lupus erythematous) or has any other disease that may be affected by immunotherapy.
* Prior treatment within 12 months of randomization with an immune modulating/immune depleting agents, such as teplizumab (TZield), thymoglobulin (ATG) or rituximab.
* Prior treatment within 6 months of randomization with a metabolic therapy intended to alter the disease course of T1D (e.g. teplizumab).
* Has significant and uncontrolled disease/condition in the investigator's opinion that may adversely affect study participation or may compromise the study results or increase participant risk.

Ages: 8 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-11-13 (Estimated); Primary Completion 2028-05-13 (Estimated); Study Completion 2029-05-13 (Estimated)

PRIMARY OUTCOMES:
The area under the stimulated C-peptide curve (AUC) Y_MAUC. | 12 Months
  The primary outcome of each participant is the mean area under the stimulated C-peptide curve (AUC) over the 2-hour mixed meal glucose tolerance test conducted at the 12-month visit in nmol/L, denoted as Y_MAUC.

SECONDARY OUTCOMES:
Effect of rezpegaldesleukin on beta cell function | From enrollment to 6 months and 12 months
  The secondary analysis will examine the effect of rezpegaldesleukin on beta cell function at 6 and 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be available at the NIDDK Central Repository
Supporting Information: Study Protocol, ICF
Time Frame: Final datasets will be available at the NIDDK Central Repository 12 months from the last participant's follow-up visit
Access Criteria: IPD can be requested through the NIDDK Central Repository once submitted.

REFERENCES:
- See also: TrialNet — http://www.diabetestrialnet.org